CLINICAL TRIAL: NCT03909152
Title: Basket Study of the Oral Progesterone Antagonist Onapristone ER (Apristor), Alone or In Combination With Anastrozole in Women With Progesterone Receptor Positive (PR+) Recurrent Granulosa Cell Tumor, Low Grade Serous Ovarian Cancer or Endometrioid Endometrial Cancer
Brief Title: A Study of Onapristone ER Alone Or In Combination With Anastrozole in Gynecologic Cancers That Respond to Progesterone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Context Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-061
Record Dates: First submitted 2019-04-08; First posted 2019-04-09 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2024-09

CONDITIONS: Granulosa Cell Ovarian Cancer; Low Grade Serous Ovarian/ Primary Peritoneal Cancer; Endometrioid Endometrial Cancer
Keywords: Onapristone ER (Apristor); Oral Progesterone; Progesterone Receptor Positive (PR+); Anastrozole; 19-061
MeSH Terms: interventions — Anastrozole

STUDY DESIGN:
Intervention Model Description: A non-randomized, open, multicenter phase 2 study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PR+ Granulosa cell tumor (This Arm is CLOSED) (Experimental): Enrolled patients will initiate treatment with onapristone ER 50 mg by mouth twice daily, about 12 hours apart, beginning Day 1 of Cycle 1. A Cycle is 28 days. This Arm is CLOSED.
  Interventions: Drug: Onapristone ER
- PR+ Low grade serous ovarian cancer (Experimental): Enrolled patients will initiate treatment with onapristone ER 50 mg by mouth twice daily, about 12 hours apart, beginning Day 1 of Cycle 1. A Cycle is 28 days
  Interventions: Drug: Onapristone ER
- PR+ Endometrioid endometrial cancer (Experimental): Enrolled patients will initiate treatment with onapristone ER 50 mg by mouth twice daily, about 12 hours apart, beginning Day 1 of Cycle 1. A Cycle is 28 days
  Interventions: Drug: Onapristone ER
- PR+ Granulosa cell ovarian cancer (Experimental): Enrolled patients will initiate treatment with onapristone ER 50 mg by mouth twice daily, about 12 hours apart and anastrozole 1mg po QD in AM beginning Day 1 of Cycle 1. A Cycle is 28 days.
  Interventions: Drug: Onapristone ER + Anastrozole

INTERVENTIONS:
Drug: Onapristone ER — 50 mg PO BID (with dosage adjustments) until POD, unacceptable toxicity or withdrawal of consent.
  Arms: PR+ Endometrioid endometrial cancer; PR+ Granulosa cell tumor (This Arm is CLOSED); PR+ Low grade serous ovarian cancer
Drug: Onapristone ER + Anastrozole — Onapristone ER Patients will take 50 PO BID in the form of two 20 mg tablets and one 10 mg tablet taken with food and water twice daily. Patients will be prescribed anastrozole 1mg PO QD. Anastrozole will be taken once daily in the AM with patients morning dose of onapristone ER.
  Arms: PR+ Granulosa cell ovarian cancer

SUMMARY:
The purpose of this study is to test any good and bad effect of the study drug, onapristone extended-release (ER) alone and in combination with anastrozole.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis at MSK of either (1) granulosa cell ovarian cancer, (2) low grade serous ovarian/ primary peritoneal cancer, or (3) endometrioid endometrial cancer; with PR expression ≥1% by IHC on archival tissue taken within the prior 3 years or new biopsy if no archival tissue is available. IHC results do not have to be from MSK.
* Measurable disease as defined by RECIST 1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension. Each lesion must be ≥10mm when measured by CT or MRI. Lymph nodes must be ≥15mm in short axis when measured by CT or MRI
* Patients must have had one prior chemotherapy regimen for management of disease. Note: additional lines of chemotherapy, biologic or immunotherapy are allowed.
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy
* At least 4 weeks out from their last dose of radiation therapy
* At least 4 weeks post-op from any major surgical procedure
* At least 3 weeks out from their last dose of chemotherapy and/or biologic/targeted therapy
* Must be ≥ 18 years of age
* Karnofsky Performance Status (KPS) of ≥ 70%
* Women of child-bearing potential must have a negative pregnancy test within 14 days prior to commencement of study treatment
* Women of child bearing potential must use an effective form of contraception during study and for at least 6 months after completion of study treatment
* Laboratory Test Findings performed within 14 days prior to initiation of study drug showing:
* Bone marrow function:

  * Absolute neutrophil count (ANC) ≥ 1,000/mcL
  * Platelets ≥ 75,000/mcL
  * Hemoglobin ≥ 8 g/dL
* Renal function:

  °Creatinine ≤ 1.5 x ULN
* Hepatic function:

  * Bilirubin ≤ 1.5 x ULN
  * AST and ALT ≤ 2.5 x ULN
* Resolution of all acute toxic effects of prior therapy to NCI CTCAE (Version 5.0) Grade ≤ 1, with the exception of unresolved Grade 2 neuropathy and Grade 2 alopecia, which are allowed
* Patient has recovered from any prior radiotherapy
* Patients must be able to swallow tablets whole, without crushing

Exclusion Criteria:

* History of another invasive malignancy (other than non-melanoma skin cancer or curatively treated in situ carcinoma) with evidence of disease within the past 3 years
* History of prior hormonal therapy (i.e., megesterol acetate, tamoxifen or aromatase inhibitors) for treatment of cancer within 28 days before starting study drug
* Any psychological, familial, sociological or geographic condition that would potentially hamper compliance with the study protocol
* Known brain metastasis which have not been treated or showed stability for ≥ 6 months
* Patient has received an oral or IV corticosteroid within the prior 28 days and requires chronic corticosteroid therapy (excludes use of steroid premeds for CT allergy)
* Uncontrolled hypertension (systolic BP ≥ 160 mmHg or diastolic BP ≥ 95mmHg) despite medical treatment. Patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment.
* Clinically significant heart disease as evidenced by myocardial infarction or arterial thrombotic event within the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class II-IV heart disease or cardiac ejection fraction measurement of < 50% at baseline
* Refractory nausea and vomiting, requirement for parenteral hydration and/or nutrition, drainage gastrostomy tube, malabsorption, external biliary shunt, or significant small bowel resection that would preclude adequate study drug absorption
* Anticipated or ongoing administration of anti-cancer therapies other than those administered in this study
* Use of any prescription medication during the prior 28 days of first onapristone dosing that the investigator judges is likely to interfere with onapristone activity; specifically strong inhibitors or inducers, or sensitive substrates of cytochrome P450 CYP3A4. Investigators should consult the following table of clinically-relevant products http://medicine.iupui.edu/CLINPHARM/ddis/clinical-table.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — GYN cancer
Enrollment: 34 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Grisham, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PR+ Granulosa Cell Tumor (This Arm is CLOSED) | PR+ Low Grade Serous Ovarian Cancer | PR+ Endometrioid Endometrial Cancer | PR+ Granulosa Cell Ovarian Cancer
Started | 14 | 5 | 1 | 14
Completed | 0 | 0 | 0 | 0
Not Completed | 14 | 5 | 1 | 14
Not completed — Adverse Event | 14 | 5 | 1 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PR+ Granulosa Cell Tumor (This Arm is CLOSED) | PR+ Low Grade Serous Ovarian Cancer | PR+ Endometrioid Endometrial Cancer | PR+ Granulosa Cell Ovarian Cancer | Total
Number analyzed (Participants) | 14 | 5 | 1 | 14 | 34
Age, Continuous [Median (Standard Deviation); unit: years] | 62.5 (29) | 59 (25) | 65 (1) | 58 (32) | 60 (24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 5 | 1 | 14 | 34
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2 | 4
  Not Hispanic or Latino | 13 | 4 | 1 | 12 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 0 | 1 | 10
  White | 8 | 0 | 0 | 11 | 19
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 5 | 1 | 14 | 34

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: as determined by RECIST 1.1 response. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = Complete Response + Partial Response (CR + PR)
Time Frame: within 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | PR+ Granulosa Cell Tumor (This Arm is CLOSED) | PR+ Low Grade Serous Ovarian Cancer | PR+ Endometrioid Endometrial Cancer | PR+ Granulosa Cell Ovarian Cancer
Number analyzed (Participants) | 14 | 5 | 1 | 14
Participants
  Participants with Overall Response Rate (Complete Response + Partial Response) | 0 | 0 | 0 | 0
  Participants with no Overall Response Rate (Complete Response + Partial Response) | 14 | 5 | 1 | 14

ADVERSE EVENTS:
Time Frame: Up to 36 weeks
Arm/Group | PR+ Granulosa Cell Tumor (This Arm is CLOSED) | PR+ Low Grade Serous Ovarian Cancer | PR+ Endometrioid Endometrial Cancer | PR+ Granulosa Cell Ovarian Cancer
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/5 | 0/1 | 0/14
Serious Adverse Events (participants affected / at risk) | 2/14 | 3/5 | 0/1 | 3/14
Other Adverse Events (participants affected / at risk) | 14/14 | 5/5 | 1/1 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PR+ Granulosa Cell Tumor (This Arm is CLOSED) (N=14) | PR+ Low Grade Serous Ovarian Cancer (N=5) | PR+ Endometrioid Endometrial Cancer (N=1) | PR+ Granulosa Cell Ovarian Cancer (N=14)
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Duodenal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PR+ Granulosa Cell Tumor (This Arm is CLOSED) (N=14) | PR+ Low Grade Serous Ovarian Cancer (N=5) | PR+ Endometrioid Endometrial Cancer (N=1) | PR+ Granulosa Cell Ovarian Cancer (N=14)
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 1 | 0 | 3
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 3
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Breast edema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0
Constipation (General disorders) | 3 | 1 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 4 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Duodenal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Edema limbs (General disorders) | 2 | 1 | 0 | 1
Fatigue (General disorders) | 5 | 0 | 0 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Hallucinations (Psychiatric disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 4
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hot flashes (Vascular disorders) | 1 | 2 | 0 | 3
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 1
Localized edema (General disorders) | 1 | 0 | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 2 | 0 | 0
Neck edema (General disorders) | 1 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 1
Paresthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 2 | 0 | 0 | 4
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1 | 0 | 1
Weight loss (Investigations) | 3 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT03909152/Prot_SAP_000.pdf